CLINICAL TRIAL: NCT03609684
Title: The Effects of Core Stabilization Exercise Program On Physical Fitness Among Amateur Artistic Gymnasts
Brief Title: Core Stabilization Exercise Program Among Amateur Artistic Gymnasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burcu Dericioğlu, Research Assistant, Eastern Mediterranean University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ETK00-2018-0156
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Therapy, Exercise; Physical Fitness
Keywords: core stabilization; endurance; gymnastics; children
MeSH Terms: conditions — Motor Activity | interventions — Gymnastics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gymnastic and Core Stabilization (Experimental): This group consist people who regularly do gymnastics and also do 30-45 minutes core stabilization exercises.
  Interventions: Other: Gymnastic and Core Stabilization
- Only Gymnastic Training (Experimental): People can do gymnastics twice a week during 8 weeks but can't do core stabilization exercise.
  Interventions: Other: Only Gymnastic Training
- Sedentary Group (Active Comparator): This group consist individuals who are not interested in any sports and don't do any exercises during 8 weeks.
  Interventions: Other: Sedentary Group

INTERVENTIONS:
Other: Gymnastic and Core Stabilization — People who regularly do gymnastics and also do 30-45 minutes core stabilization exercises
  Arms: Gymnastic and Core Stabilization
Other: Only Gymnastic Training — People can do gymnastics twice a week but can't do core stabilization exercise
  Arms: Only Gymnastic Training
Other: Sedentary Group — People who are not interested in any sports and don't do any exercises
  Arms: Sedentary Group

SUMMARY:
Purpose of this study ; to examine the effect of core stabilization program for gymnasts.The individuals has to divided into 3 groups. First group will consist individuals who are not interested in any sports and don't do any exercises during 8 weeks. Second group people can do gymnastics twice a week but can't do core stabilization exercise. Third group is consist people who regularly do gymnastics and also do 30-45 minutes core stabilization exercises as well.

DETAILED DESCRIPTION:
Core stabilization is an ability which describes the control of movements in kinetic chain during changes in positions at terminal segments . Hodges and Richard examined muscle activations during movements and found that some muscles which are responsible from core stabilization start to activate before extremity muscles.These results can support the hypothesis of movements come from control and stabilization through core. The body or as specified lumbopelvic area can contain spine cord and pelvis stabilization at work of active, passive and neutral. All these systems are work together for one purpose/Passive system contain bonds, vertebrates and invertebrates , neutral system consist nerve and central nerve system . In active system there are muscles within tendons ,core muscles can be describe as double cylinder and it's the investigator's body's power supply. This double cylinder's front consist abdominal muscles and back of it consist paraspinal muscles, above area is diaphragm and down is from pelvic and hip muscles.

Performance of muscles show the capacity of its work done.There are three important subtitles to show this performance , force , power and endurance . Especially for professional athletes if the performances are not enough or one of them can be not consist it means they effected in immortal ways. One of these elements , muscle endurance is the resistance of muscle for the stretching for a time and stay constant in this situation and show resistance ability to fatigue. This is needed to lot of activities during the day however in sport activities we need balance as top level , coordination and improve performance as an element.There is a defense which says that improvement of muscle endurance has an importance role for making stronger muscles and at the same time it is also be shown as making muscles strong. In order to make stronger muscles ACSM (American College of Sports Medicine) suggested to exercise 3 times a week by making each exercise 2-4 sets . For improvement of force and power we need to exercise up to 8-12 sets and for muscle endurance we need 15-20 repeated sets.

Gymnastics; a multidirectional sport which consist of speed , force , endurance , flexibility , agility , power and balance. If you want to be successful and make this sport as a professional you need to have suitable physical appearance and an ability. In this situation it is important to make core muscles powerful. In recent years the exercises of core stabilization has an importance role to prevent or decrease backache and also it is used as a concept of therapy for improving physical relevance and performance. It is shown in may researches that core stabilization can affect the balance to the specific movements in gymnastics as well as core endurance and if it is not enough it affect the performance in bad ways and may be increase the risk of injury.

In literature there are researches which show positive correlations between core stabilization and performance. For this reason, gymnastic coaches has to add core stabilization in their exercise list. In this care core endurance and performance which is related to balance can be directly increase. We seen that there is a lack of strengthening core stabilization program in literature. Purpose of this study ; to examine the effect of core stabilization program for gymnasts.The work consist amateur 7-9 years old children. The individuals has to divided into 3 groups. First group will consist individuals who are not interested in any sports and don't do any exercises during 8 weeks. Second group people can do gymnastics twice a week but can't do core stabilization exercise. Third group is consist people who regularly do gymnastics and also do 30-45 minutes core stabilization exercises as well.Gymnastic training is going to be given by a professional coach from Turkish Republic of Nothern Cyprus Gymnastic Federation twice a week as one hour. Generally these training consist the movements to improve the power and flexibility of individuals plus as a professional meaning which consist specific things like ; bridge , glider , eagle , spagat , circle , flick flack and perpendicular stance. It is worked for making strongest protocol core stabilization in different source of literatures. As a result they confirm of a progress in two weeks as exercising in 8 weeks. This progress consist 30-45 minutes\ day and 3 days\ week. Before every training they need to have 10 minutes warming exercises. This include 5 minutes running and 5 minutes stretching of all groups of muscles. All the exercises have to be combined with breathing.

ELIGIBILITY:
Inclusion Criteria:

* 7-9 years child gymnasts
* At least 3 months regularly attending children
* Girl children

Exclusion Criteria:

* People who has at least 6 months extremity and lack of spine surgeon
* Neurological ,vestibular and people who has vizuel problems except breakage.

Ages: 7 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — There are differences in physical and physiological between genders. These differences can effect directly to the performance. Also after puberty these differences are become evident. From infant period parents , teachers , coaches can separate boys and girls according to their physical activities which can be affect their fat ratio of body or muscle texture.This is the reason that man can be successful at short which needs force and woman can be successful at gymnastics which needs flexibility.
Enrollment: 51 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Core Endurance | Change from baseline the core endurance tests at the end of 8 weeks
  Muscle endurance is the resistance of muscle for the stretching for a time and stay constant in this situation and show resistance ability to fatigue.Body muscle endurance is going to tested by Mc Gill and his friends in 1999. The goal of the test is to look at people who stay at 3 different static positions. These tests are formed from body flexion , extension (Biering-Sorensen Test) and side bridge. When the static position continue or become up to 240 seconds the test will be ended.

SECONDARY OUTCOMES:
Static Balance | Change from baseline the static balance tests at the end of 8 weeks
  It's the ability of body which control the body at static , dynamic positions. The Flamingo balance test will be used to measure the static balance.Individuals are going to stand balanced on a wooden beam on bare feet in a position similar to flamingos. This wooden beam will be 50 cm long , 4 cm high and 3 cm wide. Stopwatch started with 'Start' command. When the balance addle stopwatch stopped and will be started when they stand on wooden beam again. About one minute they try to move. If there are more than 15 balance faults in 30 seconds the test will be ended and zero points will be given. When one minute finished the test ended and individuals faults will have calculated .
Dynamic Balance | Change from baseline the dynamic balance test at the end of 8 weeks
  In order to test dynamic balance individual's have to stay on embodiments on their dominant foot and with free foot because they need to reach to their dominant foot according to Anterior, Posteromedial and Posterolateral types. For dominant foot it is repeated 3 times up to 120 seconds. After 3 repetitions the result of this test has to be done by looking maximum number and written in cm.
Explosive Power | Change from baseline the explosive power test at the end of 8 weeks
  Explosive power is defined as the ability to produce high forces together with muscle contraction for a very short period of time. Vertical jumps will be used for evaluate the explosive power.The individuals who wants to enter the test has to stand by the wall in side position. They extend arm and get the result of longest finger. Later individuals needed to jump at highest position with a flexion position of body with knees and hip and arms have to be two-sided. The first and last handed areas are going to measured in centimeters. The jumping will be repeated 3 times and every repetition there will be 60 seconds break. After 3 jumping the best one will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Dericioğlu, Res Assist., Principal Investigator — EMU Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Emine H. Tüzün, Prof. Dr., Study Chair — EMU Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Berkiye Kırmızıgil, Assist. Prof, Principal Investigator — EMU Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Levent Eker, Assist. Prof, Principal Investigator — EMU Faculty of Health Sciences, Physiotherapy and Rehabilitation Department
Locations (2):
- Turkey (Türkiye) (2):
  - Eastern Mediterrenean University, Mersin
  - EMU Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Mersin

IPD SHARING:
Plan to Share IPD: No